CLINICAL TRIAL: NCT02619487
Title: The Impact of Mobile Technology on Clinical Outcomes in Children and Adolescents With Type 1 Diabetes
Acronym: Edu4U
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to limited staff resources, we were unable to start enrolling participants.
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Gwendolyn Pierce, Research Nurse, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 01
Record Dates: First submitted 2015-06-08; First posted 2015-12-02 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 8-12 years old, parent receiving text (Experimental): text message to parent only
  Interventions: Other: text message to parent only
- 13-18 years old, parent receiving text (Active Comparator): text message to parent only
  Interventions: Other: text message to parent only
- 13-18 years, both receiving text (Active Comparator): Text message to parent and adolescent
  Interventions: Other: text message to parent and adolescent
- No text (No Intervention): No text will be sent

INTERVENTIONS:
Other: text message to parent only — A weekly text message of an educational or motivational nature and related to Type 1 Diabetes will be sent for a duration of one year
  Other Names: e-health intervention
  Arms: 13-18 years old, parent receiving text; 8-12 years old, parent receiving text
Other: text message to parent and adolescent — A weekly text message of an educational or motivational nature and related to Type 1 Diabetes will be sent for a duration of one year
  Arms: 13-18 years, both receiving text

SUMMARY:
The purpose of this study is to determine whether a simple text message reminder sent to the parent of an child/adolescent with Type 1 Diabetes(or parent and adolescent) is effective in helping the individual(or parent) become more compliant with self-managing the Type 1 Diabetes (T1D). There will be 5 arms: text message sent to parents of children age 8-12 years old with T1D, text messages sent to parents of adolescents ,age 13-18 years old, with T1D,text messages sent to parents of adolescents with T1D as well as the adolescent with T1D,no text message sent to parents of children age 8-12 years, and no text message sent to adolescents or parents of adolescents age 13-18 years old.

DETAILED DESCRIPTION:
Managing Type 1 Diabetes requires daily checks of blood glucose and medication adjustments. Children and adolescents are known to have more difficulty with this than adults. Parents/legal guardians also face the task of helping with this self-management. A weekly text message regarding Type 1 Diabetes, sent to the parent or the parent and adolescent, may help to remind and motivate an individual to perform the daily tasks needed to manage their Type 1 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing to agree to participate(assent) in the study and have the permission of the parent to do so.
2. Have a diagnosis of Type 1 diabetes for ≥ one year.
3. Be aged 8 to 18 years old.
4. Be on insulin therapy for ≥ one year.
5. Have a parent/legal guardian with access to a working cell phone or have a parent/legal guardian with access to a working cell phone and have a working cell phone (if 13 years of age or older).
6. Utilize one of the following mobile carriers: T-Mobile, Sprint, Verizon, AT&T, or Virgin Mobile.
7. The parent/legal guardian must express intent to maintain a carrier plan for the duration of the study.
8. The parent/legal guardian must be able to read English OR the parent/legal guardian and the adolescent must be able to read English.

Exclusion Criteria:

1. Participants, who in the opinion of the investigator, have any contraindication to tight glycemic control.
2. Individuals who are unable to undertake blood glucose testing during the study period
3. Individuals who are deemed unable or unlikely to comply with the protocol.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-12-13 (Estimated); Study Completion 2019-12-13 (Estimated)

PRIMARY OUTCOMES:
glycemic control assessed by HbA1C level. | up to one year after randomization occurs
  review of lab value

SECONDARY OUTCOMES:
number of episodes of Diabetic Ketoacidosis (DKA) | up to one year after randomization occurs
  chart review of self reported episodes of Diabetic Ketoacidosis and chart review of hospitalizations related to DKA
number of episodes of severe hypoglycemia | up to one year after randomization occurs
  chart review of reported episodes of severe hypoglycemia and chart review of hospitalizations related to hypoglycemia
number of patient contacts to the diabetes educator | up to one year after randomization occurs
  chart review of educator documentation of communication with subject
number of hospitalizations related to T1D | up to one year after randomization occurs
  chart review of hospitalizations related to T1D

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn S Pierce, MSN, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No